CLINICAL TRIAL: NCT04639154
Title: Effect of Tramadol Hydrochnoride as Adjuvant to Local Anesthetic in Ultrasound Guided Erector Spinea Plane Block in Management of Chronic Chest Wall Cancer Pain: a Randomized Controlled Trial
Brief Title: Tramadol Hydrochnoride as Adjuvant to Local Anesthetic in Ultrasound Guided Erector Spinea Plane Block in Management of Chronic Chest Wall Cancer Pain
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Shereen Mamdouh, Associate professor, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 495
Record Dates: First submitted 2020-11-17; First posted 2020-11-20 (Actual); Last update posted 2021-08-03 (Actual); Status verified 2021-07

CONDITIONS: Chronic Pain; Erector Spinea Plane Block
Keywords: chronic chest pain, tramadol hydrochroide, erector spinea plane block
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control group (Placebo Comparator): patients will receive a solution of 28 ml of bupivacaine 0.25% and 2 ml of NaCl 0.9% will be added to the local anesthetic solution divided into two levels of injection T5 and T8 in ipsilateral ESPB
  Interventions: Procedure: Erector spinea plane block
- tramadol 50 (Active Comparator): patients will receive a solution of 28 ml of bupivacaine 0.25% and 2 ml of tramadol hydrochloride 50 mg will be added to the local anesthetic solution divided into two levels of injection T5 and T8 in ipsilateral ESPB.
  Interventions: Procedure: Erector spinea plane block
- tramadol 100 (Active Comparator): patients will receive a solution of 28 ml of bupivacaine 0.25% and 2 ml of tramadol hydrochloride 100 mg will be added to the local anesthetic solution divided into two levels of injection T5 and T8 in ipsilateral ESPB.
  Interventions: Procedure: Erector spinea plane block

INTERVENTIONS:
Procedure: Erector spinea plane block — ESPPB will be performed at the T5 and T8 levels of the spine using an in-plane approach. A real-time ultrasound machine will be used to evaluate block performance. A high frequency linear ultrasound probe will be placed longitudinally at a distance of 3 cm from the midline. After identifying the erector spinae muscle and transverse processes, we will insert a 22 G, 100-mm needle after standard skin disinfection. It will be inserted in a caudal-to-cephalad direction using a sterile probe cover until the tip lay in the interfacial plane deep into the erector spinae muscle. This plane will be opened following hydrolocalization with normal saline then 30 mL of 0.25% bupivacaine will be injected slowly, with or without adjuvants, and aspirate every 5 ml to ensure block performance.

SUMMARY:
Chest wall pain is a severe and distressing symptom. The erector spinae plane block (ESPB) is an interfascial plane block where local anesthetic is injected between the erector spine muscle and the transverse process. It is a simple procedure, with easy sonographic landmarks, for postoperative analgesia in patients undergoing thoracic, abdominal, lumbar, and urologic surgery. The ESPB was initially described to relieve chronic pain from metastatic disease and rib fractures.

DETAILED DESCRIPTION:
Chest wall pain is a severe and distressing symptom.Interventional pain management aims to use invasive techniques such as joint injections, nerve blocks and/or neurolysis, neuromodulation, and cement augmentation techniques to diagnose and treat pain syndromes unresponsive to conventional medical management. The erector spinae plane block (ESPB) is an interfascial plane block where local anesthetic (LA) is injected between the erector spine muscle and the transverse process. It is a simple procedure, with easy sonographic landmarks, for postoperative analgesia in patients undergoing thoracic, abdominal, lumbar, and urologic surgery. The ESPB was initially described to relieve chronic pain from metastatic disease and rib fractures.

The ESPB provides blockade of ventral and dorsal ramus from T1-2 to T8-12 with easy insertion of a catheter into the distension induced by the injectate. It is performed away from the pleura and neuraxis, with low risk of complications in these structures.To our knowledge it is the first time study to evaluate the effectiveness of tramadol hydrochloride as adjuvant to local anaesthetic in ultrasound guided ESPB in the management of chronic chest wall cancer pain. Our hypothesis is that tramadol, when added to the local anaesthetic solution injected for ESPB, may improve analgesia and decrease the opioid consumption in patients with chronic chest wall cancer pain

ELIGIBILITY:
Inclusion Criteria:

* patients with persistent chronic chest wall cancer pain (>6 months) with VAS pain score ≥ 5 on 0 to 10 scale despite of medical treatment with tramodine up to 200 mg daily

Exclusion Criteria:

* they have hypersensitivity to any of the studied drugs,
* obesity (BMI >35),
* presence of local pathology such as recurrent cancer or infection at the site of injection,
* abnormal coagulation profile,
* an abnormal liver or renal function
* unable to express their pain or
* patient refusal

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-03-30 (Estimated)

PRIMARY OUTCOMES:
changes in pain intensity measured by visual analog scale (VAS) | 10 minute after injection, every week for one month after the procedure, 2 month after the procedure
  scored from 0 to 10 where 0 = no pain and 10 = the worst pain imaginable

SECONDARY OUTCOMES:
a 7-point Likert- like verbal rating scale | every week for one month after the procedure
  extremely dissatisfied = 1, dissatisfied=2, somewhat dissatisfied=3, undecided=4, somewhat satisfied=5, satisfied=6, and extremely satisfied=7.
total analgesic requirement | every week for one month after the procedure, 2 month after the procedure
  tital amount of analgesia consumed by the patients after the procedure

CONTACTS AND LOCATIONS:
Locations (1):
- Assiut University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided